CLINICAL TRIAL: NCT02624934
Title: Clinical Predictive Value of Podocan and Wnt Pathway Regulatory Molecules on Maladaptive Left Ventricular Response in Aortic Stenosis
Brief Title: Podocan and Wnt Pathway in Left Ventricular Remodeling of Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: Bassett Healthcare (Other)
Collaborators: Baylor University (Other)
Responsible Party: Principal Investigator, Daniel Katz, Attending Physician - Cardiology, Bassett Healthcare
Other Study IDs: 2023
Record Dates: First submitted 2015-11-04; First posted 2015-12-09 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aortic stenosis is a major cause of morbidity around the world. Progressive aortic stenosis leads to cardiac hypertrophy as a compensatory response. A maladaptive response may lead to heart failure at varying degrees of severity of aortic stenosis in individual patients. The predicting factors for the occurrence of a maladaptive response are not well defined. Therefore current medical therapy for aortic stenosis is considered insufficient and may actually cause harm. The only effective therapy for severe, symptomatic aortic stenosis is aortic valve replacement. It has been found in an experimental study that Podocan determines the degree of cardiac hypertrophy in response to pressure overload via the Wnt-pathway. The possible prognostic role of secreted circulating Wnt modulators in aortic stenosis has also recently gained attention. This project will attempt to establish the prognostic role of circulatory Podocan and Wnt modulators for maladaptive left ventricular response to aortic stenosis. This may help identify patients at particular risk to develop left ventricular dysfunction with aortic stenosis and improve understanding of the mechanisms of left ventricular remodeling in aortic stenosis. Hence, this may also later act as an important background in finding more effective therapies to prevent or delay maladaptive left ventricular response in aortic stenosis.

DETAILED DESCRIPTION:
Valvular heart disease is a common clinical indication to assess patients with cardiac MRI. Cardiac MRI is comprehensive study that uses multiple imaging sequences.Cardiac MRI is indicated to image native and prosthetic aortic valves. Planimetry of the aortic valve is valuable for determination of the severity of aortic stenosis. Cardiac MRI is the most accurate and reproducible imaging modality to assess left ventricular function and mass. Left ventricular (LV) function is a primary determinant of outcomes following aortic valve replacement. LV mass is increased in severe aortic stenosis. Variations in the morphology of hypertrophy in response to aortic stenosis have been detected by cardiac MRI. Cardiac MRI is commonly used to assess aortic stenosis in the context of discordant information from alternative imaging modalities and low gradient aortic stenosis.

It is expected that 100 participants will be enrolled in the study over 24 months. This is sample size was agreed upon after discussion with the statistics team.

Patients who agree to participate will provide informed consent prior to their cardiac MRI. A 6 minute walk test to measure baseline functional status will be done after consent, preferably just prior to reporting to the MRI suite for their scheduled test. Standard cardiac MRI will be obtained. All patients having a cardiac MRI have an IV line placed as normal procedure. When the line has been placed, prior to contrast infusion (if applicable)or other medication administration, blood samples will be collected to test for circulatory Podocan and Wnt pathway molecules. Approximately 20 cc will be drawn in total. All specimens will be sent to the experimental lab of Dr. Paul Klotman at Baylor Medical Center. All of the Podocan & Wnt pathway effectory molecules assays will be completed by Dr. Klotman's lab.

The following measurements will be collected from the cardiac MRI:

LV end diastolic (ED) volume: ml LV ED index: ml/m2 LV end systolic (ES) volume: ml LV ES index: ml/m2 LV ejection fraction (EF): % LV Stroke Volume: ml LV Stroke Index: ml/m2 LV Cardiac Output: L/min LV Cardiac Index: L/min/M2 LV Mass: g LV Mass index: g/m2

At 12 months post procedure the following information will be collected from the participants' charts for endpoint analysis:

All cause mortality Cardiac mortality Hospital admissions for valvular disease related clinical events such as congestive heart failure, angina, syncope Valve replacement surgery

Patients who do undergo valve replacement surgery during the 12 month follow up period and are scheduled to undergo a post-op follow up cardiac MRI (expected to be at 9-12 months post-op) will be asked to provide additional blood samples to test for circulatory Podocan and Wnt pathway molecules at the time of the MRI.

Each participant's chart will be reviewed at the time of enrollment and the following variables will be abstracted from the medical record:

age, gender, ethnicity, Most recent Ht, Wt, BP, Heart Rate BMI Tobacco use/history Alcohol use/ history Comorbidities

* Hypertension
* Hyperlipidemia
* Diabetes
* Chronic Kidney Disease
* Cancer
* CAD

Info from previous echocardiogram:

* Ejection fraction
* Valve area
* Gradient

Info from previous cardiac cath (if done):

* Presence/absence of coronary stenosis
* Location & degree of stenosis
* Aortic valve area
* Calculation of valve area

Info from previous ECG:

* Rhythm
* Left Ventricular Hypertrophy Medications

Laboratory data:

* Lipids
* Chemistries
* Complete Blood Count
* Hemoglobin A1C
* Troponin
* B-type Natriuretic Peptide

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Scheduled for Cardiac MRI
* Patients with known aortic valve area of less than 1 cm² on echocardiogram
* Able to provide informed consent
* Ambulatory and expected to be able to complete 6 minute walk test

Exclusion Criteria:

* Other significant (moderate or severe) valvular heart disease
* Unable to complete 6 minute walk test (ex. Wheelchair bound)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with know severe aortic stenosis who are scheduled for cardiac MRI
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-10; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Podocan level | Day 1
  All patients having a cardiac MRI have an IV line placed as normal procedure. When the line has been placed, prior to contrast infusion (if applicable)or other medication administration, blood samples will be collected to test for circulatory Podocan .
Wnt Pathway molecule levels | Day 1
  All patients having a cardiac MRI have an IV line placed as normal procedure. When the line has been placed, prior to contrast infusion (if applicable)or other medication administration, blood samples will be collected to test for circulatory Wnt pathway molecules

SECONDARY OUTCOMES:
Podocan level | 18 months
  Any previously evaluated participants who go on to have aortic valve replacement surgery, will have repeat blood sampling for Podocan levels at time of 9-12 month post op assessment.
Wnt Pathway molecule levels | 18 months
  Any previously evaluated participants who go on to have aortic valve replacement surgery, will have repeat blood sampling for Wnt pathway molecule levels at time of 9-12 month post op assessment.
6 minute walk test | Day 1
  To assess whether circulatory podocan is associated with improved functional capacity of patients with AS, the relationship between circulatory podocan and a six minute walk test conducted at the time of cardiac MRI will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: D Katz, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States